CLINICAL TRIAL: NCT06743880
Title: Knowledge,attitude &practice on Human Papilloma Virus Vaccination Among Healthcare Providers and General Population
Brief Title: Knowledge, Attitude &practice on Human Papilloma Virus Vaccination Among Healthcare Providers and General Population
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelaaziz Mohamed Fathi, resident doctor at Assiut University hospital, Assiut University
Other Study IDs: KAP ON HPV vaccination
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Human Papilloma Virus (HPV) Vaccine
Keywords: Knowledge,attitude &practice
MeSH Terms: conditions — Papillomavirus Infections; Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- health care provider group: - Healthcare providers at the Gynecologic Oncology Unit have direct interactions with patients and can significantly influence their knowledge, attitudes, and decision-making regarding HPV vaccination.

SUMMARY:
* Cervical cancer is caused by persistent infection with certain strains of the human papillomavirus (HPV), which is a very common virus transmitted through sexual activity.
* HPV infections can lead to the development of precancerous lesions on the cervix, which if left untreated, can progress to invasive cervical cancer over time.
* Cervical cancer is the second most common cancer among women in Egypt, after breast cancer.
* According to the latest available data, the age-standardized incidence rate of cervical cancer in Egypt is approximately 6.3 per 100,000 women.
* However, the actual burden of cervical cancer in Egypt is likely underestimated, as many cases may go undetected or unreported, especially in rural and underserved areas.

The main objectives of this KAP study are:

1. To assess the level of knowledge about HPV and HPV vaccination among the target population.
2. To investigate the attitudes and perceptions towards HPV vaccination.
3. To identify the current practices and uptake of HPV vaccination.
4. To explore the factors influencing the knowledge, attitudes, and practices related to HPV vaccination.

DETAILED DESCRIPTION:
- Cervical cancer mortality rates in Egypt are also relatively high, with an age-standardized mortality rate of around 3.2 per 100,000 women.

Risk Factors and Epidemiology:

* The primary risk factor for cervical cancer in Egypt is persistent infection with high-risk strains of the human papillomavirus (HPV), particularly HPV 16 and 18.
* Other risk factors include early age of first sexual intercourse, multiple sexual partners, high parity, smoking, and lack of regular cervical cancer screening.
* Socioeconomic factors, such as low education levels and limited access to healthcare services, also contribute to the cervical cancer burden in Egypt.
* Cervical cancer disproportionately affects women in rural and disadvantaged areas, where screening and preventive services are less accessible.

Screening and Prevention Efforts:

* Cervical cancer screening through Pap smears or HPV testing is the primary method for early detection and prevention of the disease.
* However, cervical cancer screening coverage in Egypt remains low, with only around 10-20% of eligible women being regularly screened.
* The Egyptian Ministry of Health and Population has implemented various initiatives to improve cervical cancer screening and awareness, but more efforts are needed to reach underserved populations.
* The introduction and widespread uptake of the HPV vaccine could significantly reduce the burden of cervical cancer in Egypt, but vaccine coverage remains suboptimal.
* Cervical cancer is a significant public health concern, as it is the fourth most common cancer in women worldwide, with a high mortality rate, especially in developing countries.
* Early detection through regular cervical cancer screening (e.g., Pap smears) and treatment of precancerous lesions can effectively prevent the development of cervical cancer.

Role of the HPV Vaccine:

* The HPV vaccine is a highly effective way to prevent cervical cancer and other HPV-related diseases, such as anal, penile, and oropharyngeal cancers.
* The vaccine targets the HPV strains (primarily HPV 16 and 18) that are responsible for approximately 70% of cervical cancer cases globally.
* The HPV vaccine is recommended for both girls and boys, typically starting at 11-12 years of age, as it is most effective when administered before the onset of sexual activity and potential HPV exposure.
* Widespread HPV vaccination, coupled with regular cervical cancer screening, has the potential to significantly reduce the burden of cervical cancer worldwide.

Importance of a KAP Questionnaire in Egypt:

* In Egypt, cervical cancer is the second most common cancer among women, and HPV infection is a major risk factor.
* However, HPV vaccination rates in Egypt remain relatively low, indicating a need to better understand the factors that influence vaccination uptake in the country.
* A KAP questionnaire can provide valuable insights into:
* The level of awareness and knowledge about cervical cancer and the HPV vaccine among the Egyptian population.
* Attitudes, beliefs, and misconceptions that may be hindering or promoting HPV vaccination.
* Current vaccination practices and barriers to accessing the vaccine.
* This information can then be used to develop targeted educational campaigns, address misconceptions, and implement strategies to improve HPV vaccination coverage in Egypt.
* By understanding the KAP of HPV vaccination, policymakers and healthcare providers can work to increase cervical cancer prevention efforts and improve the overall public health outcomes in the country.

ELIGIBILITY:
Inclusion Criteria:

* 1. general population:
* Eligibility criteria:
* Age: 9-79 years old
* patients and their relatives
* Attending the Obstetrics and Gynecology, or Family Medicine clinics at Assiut University Hospital
* Recruitment strategy:
* Using a systematic random sampling method, every nth patient (based on the average patient load) will be approached and invited to participate in the study.
* The target sample size for patients is a minimum of 384 participants.

  2. Healthcare providers:
* Eligibility criteria:
* Physicians, nurses, and other healthcare workers employed in the Obstetrics and Gynecology, and Family Medicine departments at Assiut University Hospital.

Exclusion Criteria:

* -Previous HPV Vaccination:
* Exclude participants who have already received the complete HPV vaccination series, as their knowledge, attitudes, and practices may differ from those who are unvaccinated.
* The study aims to understand the KAP of the unvaccinated population, which is the primary target group for intervention.

  2-Severe Cognitive or Mental Impairment:
* Exclude participants who have severe cognitive or mental impairments that may prevent them from understanding and responding to the questionnaire accurately.
* This could include individuals with advanced dementia, severe intellectual disabilities, or acute psychiatric conditions.

  3-. Inability to Provide Informed Consent:
* Exclude participants who are unable to provide informed consent due to language barriers, literacy issues, or other factors that may compromise their ability to understand the study and its implications 4- Severe Illness or Hospitalization:
* Exclude participants who are currently hospitalized or experiencing severe illness, as their focus may be on their immediate health concerns rather than the KAP questionnaire.

Ages: 9 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Physicians, nurses, and other healthcare workers employed in the Obstetrics and Gynecology, and Family Medicine departments at Assiut University Hospital.
Sampling Method: Probability Sample
Enrollment: 323 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Knowledge about HPV | baseline
  Proportion of participants with adequate knowledge about HPV
Knowledge about HPV Vaccination | baseline
  Proportion of participants with adequate knowledge about the HPV vaccine

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Brewer NT, Fazekas KI. Predictors of HPV vaccine acceptability: a theory-informed, systematic review. Prev Med. 2007 Aug-Sep;45(2-3):107-14. doi: 10.1016/j.ypmed.2007.05.013. Epub 2007 Jun 2. PMID 17628649